CLINICAL TRIAL: NCT00829920
Title: The Effect of Treatment on Circulating Tumor Cells in Bladder Cancer Patients With Muscle-invasive or Advanced Disease
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 08-0018.cc
Record Dates: First submitted 2009-01-25; First posted 2009-01-27 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Bladder Cancer
Keywords: Bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum from patients undergoing treatment for muscle-invasive or metastatic bladder cancer who are planning for surgical bladder removal or chemotherapy will be acquired.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Bladder cancer: Patients with muscle invasive or metastatic bladder cancer who will be planning for treatment with surgery or chemotherapy.

SUMMARY:
The investigators hypothesize that circulating tumor cells (CTC) will be observed in patients with muscle-invasive or metastatic bladder cancer and that CTC will become undetectable, at least transiently, in a fraction of patients after treatment. To investigate this hypothesis, investigators will assess the levels of CTCs both before and after treatment. The feasibility and potential value of fluorescent in situ hybridization (FISH) in the CTCs will be assessed.

DETAILED DESCRIPTION:
The measurement of circulating tumor cells is pursued in several cancers including breast and prostate cancer. The number of cells measured in these cancers has been shown to be prognostic. There is little information on the presence or importance of circulating tumor cells in bladder cancer. This trial is designed to determine if patients with advanced bladder cancer have circulating tumor cells and if these circulating cells are affected by treatment of the cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of transitional cell carcinoma of the urothelium of at least T2-4, Nx, Mx stage. Mixed histologies will be allowed (e.g. squamous differentiation) as long as a transitional cell component is present.
* Clinical plans for surgery (with or without chemotherapy), radiation therapy, or chemotherapy.
* Participants must not have any condition which in the investigator's opinion may compromise the feasibility of completing the study.
* Subject must be 18 years of age or older
* Subject must be willing to have up to 4 peripheral blood samples obtained over a 6 month period of study.
* Prior therapies for bladder cancer will be allowed if patient currently has muscle-invasive or metastatic bladder cancer despite the previous treatments.
* Predicted life expectancy of > 12 weeks.

Exclusion Criteria:

* Subjects who are unwilling or unable to comply with the study guidelines as determined by the principal investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with muscle-invasive or metastatic bladder cancer with plans for cancer treatment.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2008-11; Primary Completion 2012-11 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Effect of therapy | baseline and then every 2 months
  To determine the effect of therapy (cystectomy or chemotherapy) on circulating tumor cell (CTC) levels in bladder cancer patients.

SECONDARY OUTCOMES:
Presence of baseline CTC | baseline and then every 2 months
  Assess for the presence of baseline CTC in bladder cancer patients with muscle-invasive or metastatic disease.
Assessing insulin like growth factor | baseline and then every 2 months
  Determine the feasibility of assessing insulin like growth factor (IGF) I-R and c-Met by FISH in circulating tumor cells of patients with advanced bladder cancer.
Correlation between CTC levels and clinical outcome | baseline and then every 2 months
  Evaluate for any potential correlation between CTC levels and clinical outcome

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W. Flaig, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States